CLINICAL TRIAL: NCT02801643
Title: The Impact of Reward-induced Dopamine Release on Functional Connectivity: a Combined PET/fMRI Study
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, David Hsu, Assistant Professor of Psychiatry, Stony Brook University
Other Study IDs: PET/MR Pilot
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: PET; dopamine; fMRI; reward

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study would be the first to investigate the relationship between reward- and or social stimuli-induced dopamine (DA) release and neural function using a combined PET/fMRI approach. Data from this project conducted in healthy subjects will provide preliminary data for a larger grant application to study patient populations with known abnormalities in DA including schizophrenia, major depressive, substance use, and eating disorders.

DETAILED DESCRIPTION:
Aim 1. To test the relationship between reward-induced dopamine (DA) release on changes in resting state functional connectivity (RSFC) in healthy subjects. In 20 healthy adults, the investigators will examine DA release (measured using positron emission tomography, PET) in the ventral striatum, thalamus, and prefrontal cortex, as previously described. Before and after the task the investigators will examine RSFC (measured using functional magnetic resonance imaging, fMRI) between these structures, which have been shown to form functional pathways serving motivation and emotion regulation in rodents and nonhuman primates. The investigators hypothesize that DA release will impact the functional relationship between these and other structures as determined by changes in RSFC.

Aim 2. To examine the relationship between dopamine release and the Reward Positivity (RewP) potential. Subjects will be presented with the option to participate in an event-related potential (ERP) study. The investigators will correlate the amount of DA release with the amplitude of the RewP potential, an ERP that is enhanced in reward versus non-reward circumstances. Based on previous studies, the investigators hypothesize that RewP amplitude will positively correlate with dopamine release in the nucleus accumbens.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women age 18-45 who have the capacity to consent to the protocol.
2. Ability to understand and follow instructions and oriented to name, time, and place.
3. A negative urine pregnancy and toxicology screen
4. Willingness to abstain from using aspirin, NSAIDs, or anticoagulants during the study

Exclusion Criteria:

1. Left-handed or ambidextrous
2. History of seizures
3. History of strokes
4. Clinically significant, uncontrolled liver, kidney, cardiac, or pulmonary disease
5. Terminal medical diagnosis consistent with survival < 1 year
6. Serious mental impairment. Mini mental state exam of < 23/30
7. Current or past DSM-IV Axis I or neurologic disorders
8. Actively abusing substances, including alcohol (regular alcohol use during the past 6 months equal to or greater than 16 cans of beer per week or equivalent; use of street drugs or regular tobacco use during the past 6 months)
9. Unstable medical condition (≥ 3 months), or serious medical illnesses during the past three months (e.g., serious infections)
10. Unexplained loss of consciousness; history of traumatic brain injury involving loss of consciousness greater than 2 minutes
11. Currently pregnant or breastfeeding, sexually active and of child-bearing potential and not using adequate contraceptive methods
12. Childbirth or miscarriage during past 6 months, breastfeeding within 6 months of recruitment
13. Allergic to latex and/or study pharmaceuticals
14. Diabetes and/or unable to fast for up to 7 hours
15. Unable to lie comfortably in the scanner for up to 4 consecutive hours
16. Would receive a total of over 5 rems to a radiosensitive organ (bone marrow, gonads, lens of the eye) or 15 rems to any other organ or to the body as a whole during a 12 month period
17. Contraindications for MRI including neurostimulators, implanted medical devices, metal in the body, claustrophobia, weight over 440 pounds, and girth size incompatible for scanner bore.
18. Participation in a similar Social Feedback Task within 2 months of the start of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 subjects (ages 18-45 years) will be included. Male and female representation will be about equal. No ethnic/racial/gender group is excluded.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dopamine receptor binding potential | 1-3 weeks
  changes in dopamine receptor binding potential will be measured during and after a reward task or social stimulus task
Resting state fMRI | 1-3 weeks
  Resting state functional connectivity will be measured using fMRI
Event-related potential (ERP) during reward | 1-3 weeks
  ERP during a reward task is measured

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No